CLINICAL TRIAL: NCT05318378
Title: Inverting Grayscale in Conventional Orthopedics X-rays Improves Detection of Proximal Femur Fracture Among Undergraduate Medical Students
Brief Title: Inverting Grayscale Improves Detection of Proximal Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de l'arthrose, Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: BIXAM
Record Dates: First submitted 2022-03-30; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We built two series of images. Series one was composed of separated conventional and inverted images. Series two consisted of inverted and conventional X-rays of the same subject (BIXAM) shown together (Figure). An independent assessor randomly duplicated four and two images for series one and two, respectively, to evaluate the intra-observer agreement. The same assessor randomized the images' order of appearance for the two series with a free online available list randomizer (www.randomizer.org). The principal investigator was blinded to the randomization during the sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- student (Experimental): Twenty fifth-year medical students were asked to participate in the study
  Interventions: Diagnostic Test: BIXAM
- senior surgeon (Active Comparator): As controls, we asked 3 independent board-certified orthopedic surgeons to participate in the study following the same conditions as described previously.
  Interventions: Diagnostic Test: BIXAM

INTERVENTIONS:
Diagnostic Test: BIXAM — Series two consisted of inverted and conventional X-rays of the same subject (BIXAM) shown together

SUMMARY:
Proximal femur fractures (PFF) are a worldwide public health concern. A delay in the diagnosis and treatment worsens the prognosis. Inversion of grayscale is a tool available on most X-rays visualization software, and its use has been suggested to improve radiological diagnosis. The study aims to determine if using inverted grayscale radiography results in better diagnoses of PFF among medical students.

Material and Methods. The investigators evaluated the detection of PFF by fifth-year medical students on a series of 30 pelvis X-rays. The series was composed of 20 X-rays with PFF and 10 X-rays without fracture. A first reading session was set up where X-rays were presented separately in conventional and inverted grayscale. A second session one month later showed both grayscale visualizations together (BIcontrast X-rays Analysis Method - BIXAM). X-rays' order of appearance was randomized. The investigators performed the same evaluation on senior orthopedic surgeons as a control. Finally, sensitivity, specificity, and accuracy were assessed for each method (conventional, inverted, and BIXAM) with the McNemar test. Subgroup analyses were performed on the fracture localization (femoral neck, trochanteric).

ELIGIBILITY:
Inclusion Criteria:

* fifth-year medical students

Exclusion Criteria:

* other medical students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
accuracy | one month
  accuracy was compared between conventional and inverted grayscales or both images shown together (BIXAM series) with non-parametric McNemar test
Sensibility, specificity, | one month
  Sensibility, specificity were compared between conventional and inverted grayscales or both images shown together (BIXAM series) with non-parametric McNemar test

CONTACTS AND LOCATIONS:
Overall Officials: cedric maillot, Study Director — APHP
Locations (1):
- Aphp, Paris, France

IPD SHARING:
Plan to Share IPD: No